CLINICAL TRIAL: NCT06432296
Title: A Randomized, Controlled, Multi-Center Phase III Clinical Study to Evaluate the Efficacy and Safety of M701 for Intraperitoneal Injection in Patients With Malignant Ascites Caused by Advanced Epithelial Solid Tumors
Brief Title: Treatment of Malignant Ascites Caused by Advanced Epithelial Solid Tumors With M701 Bispecific Antibody
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M70104
Record Dates: First submitted 2024-05-18; First posted 2024-05-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Malignant Ascites
MeSH Terms: interventions — Paracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- M701 group (Experimental): M701 will be administered via intra-peritoneal infusion following sufficient drainage of malignant ascites.
  The treatment regimen consists of a leading dose of 50μg on Day 1, followed by three infusions of the full dose of 400 μg M701 on Days 4, 11, and 18. If well tolerated, patients will continue to receive M701 infusions every 2 weeks as maintenance treatment.Additionally, these patients will receive systemic therapy as determined by the investigator.
  Interventions: Drug: M701
- Control group (Active Comparator): Patients in the control group will undergo paracentesis on Day 1 and Day 18. If necessary, they may receive additional paracentesis during this period. Additionally, these patients will receive systemic therapy as determined by the investigator.
  Interventions: Procedure: paracentesis

INTERVENTIONS:
Drug: M701 — Intra-peritoneal infusion of M701 in experimental group (M701 group_
  Arms: M701 group
Procedure: paracentesis — Puncture and Draiange of ascites from the peritoneal cavity in both experimental group and control group
  Arms: Control group

SUMMARY:
A Randomized, Controlled, Multi-Center Phase III Clinical Study to Compare the Efficacy and Safety of Recombinant Anti-EpCAM and Anti-CD3 Human-Mouse Chimeric Bispecific Antibody (M701) for Intraperitoneal Injection to Paracentesis alone in Patients with Malignant Ascites Caused by Advanced Epithelial Solid Tumors.

DETAILED DESCRIPTION:
The phase III study is a controlled, open-label trial designed to assess the effectiveness and safety of M701 intra-peritoneal infusion for controlling malignant ascites in patients with Malignant Ascites Caused by Advanced Epithelial Solid Tumors who are also receiving systemic therapy.

A total of 270 patients with malignant ascites caused by Malignant Ascites Caused by Advanced Epithelial Solid Tumors will be randomly assigned to two treatment arms in a 2:1 ratio. These patients must have experienced disease progression or intolerance after receiving at least two lines of systemic therapy.

Both treatment arms will receive the systemic therapy as per the investigator's instructions. The test arm will receive paracentesis and intra-peritoneal infusion of M701, while the control arm will receive paracentesis alone.

The primary endpoint of the study is the puncture-free survival, which evaluates the efficacy of M701 in controlling malignant ascites. Secondary endpoints include the overall survival (OS),Time to next puncture (TTNP), Patient-reported outcome (PRO) score, 6-month survival rate,1-month and 2-month puncture-free survival rate, safety profiles,and Anti-m701 antibody (ADA) and Neutralizing antibody (NAb).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign the written informed consent form;
2. Age ≥18 years and ≤75 years;
3. Histologically or pathologically confirmed epithelial malignant solid tumors,including: advanced gastric cancer and colorectal cancer that have failed at least two lines of treatment (treatment failure is defined as progression after treatment or intolerance after treatment); or platinum-resistant (platinum-efractory) dvanced ovarian cancer;
4. Pathologically or clinically diagnosed with malignant ascites, and treatment for malignant ascites is required as judged by the investigator; B-mode ultrasound confirms that the volume of ascites is moderate or above (moderate or above ascites is defined as the maximum depth of ascites by B-mode ultrasound in supine position is ≥ 4.5 cm, or the actual amount of ascites drained is ≥ 1 L;
5. The time interval between the last anti-tumor treatment and Randomization should meet the following time intervals:

   1. Intraperitoneal therapy: The time from the most recent intraperitoneal infusion therapy to randomization should be ≥ 2 weeks;
   2. Systemic treatment: No washout required;
   3. AEs should have recovered to Grade ≤ 1 from previous treatment (except for other adverse reactions (such as alopecia) that do not affect the safety evaluation of the investigational drug as judged by the investigator according to NCI-CTCAE V5.0);
6. ECOG PS score of 0 to 2;
7. An expected survival of ≥ 8 weeks;
8. Organ functions must meet the following criteria:

   1. Hematology: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelets ≥90 ×10^9/L, hemoglobin ≥ 85 g/L, and lymphocyte percentage ≥ 10%;
   2. Liver function: total bilirubin ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN (AST and ALT ≤ 5 × ULN are allowed in case of liver metastasis);
   3. Serum albumin ≥ 28 g/L;
   4. Renal function: serum creatinine ≤ 1.5 × ULN.
9. Female subjects of childbearing potential should have a negative pregnancy test at screening; all female subjects of childbearing potential and male subjects should take adequate contraceptive measures throughout the treatment period and within 6 months after the end of the study.

Exclusion Criteria:

1. Patients with a known history of allergy to M701 or its components; patients with a known history of allergy to macromolecular ntibody drugs or a history of specific allergic reactions (asthma, rubella, and eczematous dermatitis);
2. Have previously used M701, or have used antibody drugs targeting EpCAM and/or CD3 within 4 months before the first dose;
3. Patients with central nervous system (CNS) metastases resulting in clinical symptoms or requiring therapeutic intervention; patients with previously treated brain metastases can be enrolled if they are asymptomatic and have stable disease as indicated by imaging examination ≥ 4 weeks before the first dose and do not require corticosteroids or anticonvulsant therapy;
4. Have undergone major surgery within 4 weeks prior to randomization or plan to undergo major surgery during the study(excluding exploratory surgery);
5. New or concurrent infection within 14 days prior to randomization that has not been controlled to clinical stability;
6. Patients with severe respiratory diseases at screening, leading to respiratory failure or those judged by the investigator to be unsuitable for enrollment;
7. Patients with active autoimmune diseases (e.g., inflammatory bowel disease,idiopathic thrombocytopenic purpura, lupus rythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, and rheumatoid arthritis), but patients with the following conditions are allowed to be screened: type I diabetes;hypothyroidism that can be controlled by replacement therapy only; skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, and alopecia);
8. Patients with severe cardiovascular and cerebrovascular diseases at screening,including cardiac insufficiency (NYHA Class III-IV); acute cardiovascular and cerebrovascular events (acute myocardial infarction, acute cerebral infarction,unstable angina, cerebral hemorrhage, etc.) orundergone vascular stenting within 6 months(Coronary artery stent implantation, intracranial artery stent implantation,etc.) or pulmonary embolism within the past 6 months; or venous thrombotic diseases such as venous thrombosis in lower limb within the past month;
9. Patients with complete intestinal obstruction within 30 days prior to Randomization,or those diagnosed with subileus but judged by the investigator as unsuitable for participating in the study based on their symptoms, signs, etc., or those have severe gastrointestinal disease such as gastric/intestinal perforation;
10. Unable to drain the ascites completely due to objective reasons (including ascites septation) or complicated with chylous ascites;
11. Portal vein embolism or portal hypertension confirmed by examinations;
12. Patients with active chronic hepatitis B [such as positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis B core antibody (HBcAb), and HBV DNA ≥2000 IU/mL or HBV DNA ≥5000cps/mL], active hepatitis C [such as positive hepatitis C virus (HCV) antibody and HCV RNA ≥ lower limit of detection], positive human immunodeficiency virus (HIV) antibody, or active syphilis infection (positive syphilis-specific antibody and positive syphilis non-specific antibody);
13. Patients with concurrent pleural effusion and clinical symptoms such as chest tightness and dyspnea, who have received clinical intervention or require clinical intervention as assessed by the investigator; or those with concurrent moderate to severe symptomatic pericardial effusion;
14. Pregnant or lactating women;
15. History of definitive neurological or mental disorders that, per the investigator's judgment, may affect the cognitive function or compliance of the patient, including unstable epilepsy, dementia, and schizophrenia;
16. Other conditions that the investigator considers unsuitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
PuFS | Time from the end of drainage of C1V4 ascites to the start of the next drainage or death (up to 6 months).
  Defined as the time from the end of C1V4 ascites drainage to the next drainage (based on the time of puncture) or the time of death is recorded as the PuFS.

SECONDARY OUTCOMES:
OS | Time from randomization to death from any cause (up to 6 months).
  Time from randomization to death from any cause

OTHER OUTCOMES:
TTNP | Time from the end of drainage of C1V4 ascites to the beginning of the next drainage (up to 6 months).
  Time from the end of drainage of C1V4 ascites to the beginning of the next drainage (as the time of drainage)
The score of quality of life | Time from randomization to end of treatment. (up to 6 months).
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 V3.0) was used to evaluate the quality of life of the subjects. This questionnaire is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients. For the first 28 questions, the score is from 1-4, the lower score represents the better quality. For the last 2 quesionts, the score is from 1-7, the higher score represents the better health and quality of life.
1-month and 2-month PuFS rates | 1st and 2nd month from randomization
  1-month and 2-month PuFS rates
6-month survival rate | 6th month from randomization
  6-month survival rate
Indidence of Adverse events | From the time of first dosing (Day 1) until one month after the end of treatment
  Incidence of Treatment-Emergent Adverse Events, ≥grade 3 Treatment-Emergent Adverse Events, Serious Adverse Events and Treatment-Related Adverse Events.
Positive rate of ADA and Nab in serum | Time from screening to end of treatment (up to 6 months).
  The positive rate of Anti-Drug Antibody (ADA) and Neutralizing antibody (Nab) in the serum during the study
The EpCAM expression in ascites | From the time of first dosing (Day 1) until the end of treatment (up to 6 months).
  Measure the count of EpCAM postive cells in the ascites before and after M701 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Xu, MD, Principal Investigator — The First Medical Center of Chinese PLA General Hospital; Yanqiao zhang, PhD, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (2):
- China (2):
  - The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang

IPD SHARING:
Plan to Share IPD: No